CLINICAL TRIAL: NCT01319227
Title: Periprosthetic Bone Remodeling Around Two Different Types of Uncemented Femoral Stems and Two Uncemented Acetabular Components in Total Hip Arthroplasty
Brief Title: Periprosthetic Bone Remodeling Around Uncemented Components in Total Hip Arthroplasty
Acronym: PeriBRUSBRAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: Johnson & Johnson Consumer Products Company Division of Johnson & Johnson Consumer Companies, Inc. (Industry)
Responsible Party: Principal Investigator, Olof Skoldenberg, Consultant Orthopaedic Surgeon, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PeriBRUSBRAC
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
Keywords: Periprosthetic bone remodeling; Stress shielding; Short femoral stem; Porous Titanium Construct; Polyethylene wear
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hip Arthroplasty, ultra-short stem, conventional cup (Experimental): Hip replacement with a hydroxy-apatite covered ultra-short uncemented femoral stem and a conventional uncemented acetabular cup with hydroxy-apatite covered porous coating and a moderately cross-linked polyethylene cup liner
  Interventions: Procedure: Hip replacement
- Hip Arthroplasty, conventional stem, trabecular-titanium cup (Experimental): Hip replacement with an uncemented tapered femoral stem and an uncemented acetabular cup with trabecular-Titanium backside and E-vitamin-treated polyethylene cup liner
  Interventions: Procedure: Hip replacement

INTERVENTIONS:
Procedure: Hip replacement — Hip arthroplasty with uncemented components
  Other Names: Ultra-short hydroxyapatite-coated Proxima stem and hydroxyapatite covered porous coated Pinnacle cup from DePuy, Johnson&Johnson.; Tapered, proximally porous and hydroxyapatite-coated, Bimetric stem and a Regenerex cup with trabecular-Titanium-backside from Biomet.

SUMMARY:
This is a randomized clinical trial comparing two different uncemented femoral stems and two different uncemented sockets using Dual-energy x-ray absorptiometry, Radiostereometry and clinical evaluation.

Hypothesis:

1. A short uncemented stem gives less periprosthetic bone resorption in the proximal femur than a conventional uncemented stem.
2. An uncemented acetabular component with a backside of three-dimensional Titanium porous construct gives less periprosthetic bone resorption than a backside covered with a conventional porous coating with Titanium-beads and a hydroxy-apatite layer.

DETAILED DESCRIPTION:
Consecutive patients 40-70 years old who are being planned for Total Hip Arthroplasty (THA) will be eligible for inclusion in the study.

Periprosthetic bone remodeling, migration of the components and clinical scores will be recorded prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-70 years old
2. Primary osteoarthritis of the hip
3. Type A or B femur according to Dorr10
4. Femoral anatomy allowing implantation of both femoral stems
5. Willingness and ability to follow study-protocol -

Exclusion Criteria:

1. Inflammatory arthritis
2. Abnormal femoral anatomy after hip dysplasia, not suitable for implantation of components
3. Treatment with bisphosphonates, cortisol or cytostatic drugs 6 months prior to surgery
4. Ongoing oestrogen treatment
5. Type C femur according to Dorr
6. Not suited for the study for other reason (surgeons preference)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-10; Primary Completion 2013-08 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Bone remodelling, i e change in bone mineral density around the stem, as measured with dual energy x-ray absorptiometry (DEXA) | bone mineral density (BMD) measured postoperatively at 2 years.
Bone remodelling, i e change in bone mineral density behind the acetabular component, as measured with dual energy x-ray absorptiometry (DEXA) | bone mineral density (BMD) measured postoperatively at 2 years

SECONDARY OUTCOMES:
Migration of stem components in six degrees of freedom and maximum total point motion measured with radiostereometric analysis (RSA) | at 2 years
Migration of acetabular components in six degrees of freedom and maximum total point motion of the head center measured with radiostereometric analysis (RSA) | at 2 years
Migration of acetabular components in six degrees of freedom and maximum total point motion of the head center measured with radiostereometric analysis (RSA) | at 6 and 10 years
Bone remodelling, i e change in bone mineral density around the stem and cup, as measured with dual energy x-ray absorptiometry (DEXA) | at 6 and 10 years.

OTHER OUTCOMES:
Clinical outcome measures with validated scores comparing patients receiving different stems and acetabular components | Self administred validated score outcome measures after 6 weeks, after 3, 6, 12, 24 months and after 6 and 10 years
  Validated scores included are Harris Hip Score (HHS), Euroqol 5-dimension (Eq5d) and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Department, Danderyd Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Axenhus M, Salemyr M, Mukka S, Magneli M, Skoldenberg O. Long-term evaluation of periprosthetic bone changes in ultra-short versus conventional stems in total hip arthroplasty: a 10-year follow-up of a randomised controlled trial. Hip Int. 2025 Dec 18:11207000251371283. doi: 10.1177/11207000251371283. Online ahead of print. PMID 41410176